CLINICAL TRIAL: NCT02642900
Title: Photodynamic Therapy Against Candida Spp. in Complete Denture Wearers: a Randomized Clinical Trial
Brief Title: Photodynamic Therapy Against Candida Spp. in Complete Denture Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Regina Tamaki, Professora Doutora, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DML01
Record Dates: First submitted 2015-10-07; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Photochemotherapy Reaction
Keywords: Complete denture; Candida spp; Photodynamic therapy
MeSH Terms: interventions — Photochemotherapy; Nystatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nystatin 100.000 units (Experimental): Patients were treated with a topical antifungal nystatin oral suspension(1000.000 units) 5mL every six hours/14 days. Patients were instructed to rinse the solution for 5 minutes and then to spit the solution out. Samples were collected on days 7, 14 and 30 after the end of treatment (follow-up).
  Interventions: Drug: Nystatin 100.000 units
- Photodynamic Therapy (Active Comparator): Patients used mouthwash with methylene blue 0.005% for 20 minutes (pre-irradiation time). The palatal mucosa was irradiated using a low level laser with the following settings: wavelength of 660 nm, energy density of 120 J/cm ², output power of 40 milliwatt, 2 minutes per point. PDT was performed in two sessions (one session per week). Samples were collected immediately after each clinical procedure and 30 days after the second procedure (follow-up).
  Interventions: Procedure: Photodynamic Therapy

INTERVENTIONS:
Procedure: Photodynamic Therapy — evaluate the effectiveness of photodynamic therapy (PDT) in the treatment of denture stomatitis in complete denture wearers.
  Other Names: photochemotherapy
  Arms: Photodynamic Therapy
Drug: Nystatin 100.000 units — Control group treated with nystatin
  Other Names: Nystatin
  Arms: Nystatin 100.000 units

SUMMARY:
Candida albicans is the most prevalent species in denture-related stomatitis (DS). There are several treatment options for this condition, including the use of antifungal agents such as nystatin and miconazole. The side effects and the increasing number of resistant species caused by the use of these drugs encourage the development of alternative therapies. Photodynamic Therapy (PDT) has been used as a promising treatment of stomatitis. In this randomized clinical trial, the effectiveness of PDT was evaluated. Patients in this study were allocated to two groups. One group was treated with nystatin, and the other group was treated with PDT.

DETAILED DESCRIPTION:
Different Candida species, including albicans, tropicalis, and parapsilosis, are present in the human oral microbiota, gastrointestinal tract and vagina. These species are typically harmless commensals. Candida albicans, the most prevalent species, may be present in up to 80% of healthy individuals. This species is found with high frequency in dental prostheses and is thought to be the main pathogen associated with stomatitis in elderly denture wearers. Biofilms of Candida albicans are usually found in intravenous catheters, prostheses, and these biofilms promote a high resistance to antifungal drugs. The standard treatment of stomatitis is topical antifungal agents, including nystatin and miconazole. The use of topical antifungal agents has caused some problems. Poor responses to these agents are the result of dilution and fast elimination of the drug because of the action of the saliva, which reduced the drug's concentration. The drug's toxicity can cause mild and transient gastrointestinal side effects, such as nausea, vomiting and diarrhea. Alternative treatments or adjuvant treatments have been used to treat these diseases, such as the use of probiotic bacteria and photodynamic therapy (PDT) using a non-toxic dye (photosensitizer - PS) in combination with a source of visible light with a peak wavelength suitable for absorption by the PS. The photodynamic process rapidly generates reactive oxygen species (ROS) such as peroxides, hydroxyl radicals, superoxide ions and singlet oxygen. Singlet oxygen has been implicated as the major causative agent of cellular damage in the photodynamic process, but it does not cause cellular damage in host tissues. The amount of ROS formation is the main predictor of yeast killing.

This study aimed to evaluate the effectiveness of photodynamic therapy (PDT) in the treatment of denture stomatitis in complete denture wearers.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting denture-related stomatitis, confirmed by clinical and microbiological evaluation

Exclusion Criteria:

* were based on the patients' medical history, and were excluded patients with a history of head and neck cancer, those with type III DS (classification proposed by Newton), and individuals who had received or were receiving treatment with antibiotics, antifungal agents or steroids for the past three months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Treatment evolution of participants with Candida-related denture stomatitis, treated with PDT or Nystatin, by numbers of colony forming units per milliliter (cfu/mL) recovered from the palatal mucosa, from baseline to end of treatment | through study completion, an average of 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Regina Tamaki, Profa. Dra., Principal Investigator — Associated Professor
Locations (1):
- Faculdade de Odontologia da Universidade de São Paulo, São Paulo, São Paulo, Brazil